CLINICAL TRIAL: NCT00279630
Title: Phase 1 Study on Effectiveness of Exercise on Function, Quality of Life and Disability in Patients With Posterior Tibial Tendon Dysfunction
Brief Title: Exercise and Shoe Orthoses in Treatment of Posterior Tibial Tendon Dysfunction
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University of Southern California (Other)
Responsible Party: Principal Investigator, Kornelia Kulig, Professor, University of Southern California
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 022051
Record Dates: First submitted 2006-01-17; First posted 2006-01-19 (Estimated); Last update posted 2014-12-03 (Estimated); Status verified 2014-12

CONDITIONS: Tendinopathy
Keywords: Tibialis Posterior Tendinopathy
MeSH Terms: conditions — Tendinopathy | interventions — Orthotic Devices; Exercise

STUDY DESIGN:
Who Masked: Outcomes Assessor

ARMS (1):
- type of exericse (Experimental): type of exercise
  Interventions: Procedure: Orthoses and Exercise

INTERVENTIONS:
Procedure: Orthoses and Exercise — orthrose and exercise - daily

SUMMARY:
Posterior tibial tendon dysfunction (PTTD) is the most common cause of painful and debilitating acquired flatfoot deformity in adults. The dysfunction is often progressive and may result in attenuation of the PTT and eventually collapse of the plantar arch or even rupture of the tendon. Current therapeutic management of PTTD is multipronged and includes management with foot orthoses, stretching, and strengthening exercises. Evidence drawn from research related to the management of painful chronic Achilles tendinosis suggests that eccentric strengthening of the posterior tibialis may lead to superior results compared to concentric. The purpose of this research is to determine the effectiveness of treatment interventions used in the management of PTTD.

DETAILED DESCRIPTION:
All study participants receive a pair of custom made orthoses and perform daily calf-stretches. In addition to the orthoses two groups will perform tibialis posterior specific exercises; one as concentric and the second as eccentric activation. Intervention will last 12 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Pain (> 3 months duration)
* Pain localized to the medial ankle and foot
* Swelling at the medial ankle
* Able to perform a single controlled heel lowering

Exclusion Criteria:

* Bilateral posterior tibial tendon dysfunction
* Fixed foot deformities
* Previous foot surgery
* Presence of any other concurrent foot pathology besides posterior tibial tendon dysfunction
* Ability to walk only with assistive device
* Neurological disorders
* Cognitive dysfunction
* Uncontrolled cardiovascular disease
* Evidence of cord compression
* Uncontrolled hypertension
* Infection
* Severe respiratory disease
* Pregnancy
* Current or recent history of low back pain
* Known rheumatic joint disease
* Peripheral vascular disease with sensory loss of the foot.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 45 (Actual)
Dates: Start 2002-06; Primary Completion 2014-12 (Actual); Study Completion 2014-12 (Actual)

PRIMARY OUTCOMES:
Foot Function Index; SF-36; walking distance in 5 minutes; time walking 50-ft; pain following the functional tests | pre- post- 6-month post

CONTACTS AND LOCATIONS:
Overall Officials: Kornelia Kulig, PhD, PT, Principal Investigator — University of Southern California
Locations (1):
- Department of Biokinesiology and Physical Therapy, Los Angeles, California, United States

REFERENCES:
- [Derived] Kulig K, Pomrantz AB, Burnfield JM, Reischl SF, Mais-Requejo S, Thordarson DB, Smith RW. Non-operative management of posterior tibialis tendon dysfunction: design of a randomized clinical trial [NCT00279630]. BMC Musculoskelet Disord. 2006 Jun 6;7:49. doi: 10.1186/1471-2474-7-49. PMID 16756656